CLINICAL TRIAL: NCT07309588
Title: Hyposalivation Treatment With Non-crosslinked Hyaluronic Acid and Amino Acids Solution
Brief Title: Hyaluronic Acid in the Treatment of Hyposalivation
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMS-Hyposalivation-2025-01
Record Dates: First submitted 2025-11-19; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-10

CONDITIONS: Xerostomia Due to Hyposecretion of Salivary Gland
Keywords: hyaluronic acid; amino acids; dry mouth
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: Clinical investigation for new indication of medical device. In this protocol the investigators use medical device class III, not a registerd drug.
  Study Model: Interventional, Open-label, Controlled
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group with intervention of Sunecos-200; injectable HA and AA solution (Experimental): 50 patients (age 38-78) with hyposalivation and syptoms of dry mouth were randomly selected, and the treatment protocol was applied. Exclusion criteria: smoking, pregnancy, breast feeding, diabetes, immunosuppressive treatment and neoplastic diseases. Sjögren disease and active inflammation in the oral cavity were also ruled out.
  In the study group Sunecos-200; HA and AAs solution were used as an intervention four times in 2 weeks intervals. At the beginning (qualification visit) and the end of study (2 weeks after the last intervention) the patients completed auctorial questionnaire. The pain level was measured with VAS scale. Patients also completed ( on the qualification and final visit) intraoral examination, including a "mirror test" to evaluate unstimulated saliva flow. To evaluate both unstimulated and stimulated saliva characteristic, a Saliva-Check Buffer GC test kit was used.
  Patients were asked to not change hygienic protocol and not use a saliva stimulants.
  Interventions: Combination Product: Sunecos-200 Injectable Hyaluronic acid and amino acids solution
- Control group without intervention (No Intervention): 50 patients (age 38-78) with hyposalivation and syptoms of dry mouth were randomly selected as a control group. Exclusion criteria: smoking, pregnancy, breast feeding, diabetes, immunosuppressive treatment and neoplastic diseases. Sjögren disease and active inflammation in the oral cavity were also ruled out.At the beginning (qualification visit) and the end of study (2 weeks after the last intervention in study group with intervention) the patients completed auctorial questionnaire. The pain level was measured with VAS scale. Patients also completed (on the qualification and final visit) intraoral examination, including a "mirror test" to evaluate unstimulated saliva flow. To evaluate both unstimulated and stimulated saliva characteristic, a Saliva-Check Buffer GC test kit was used.
  Patients were asked to not change hygienic protocol and discontinue the use of saliva stimulants.

INTERVENTIONS:
Combination Product: Sunecos-200 Injectable Hyaluronic acid and amino acids solution — In the study group with intervention a total of 2 mL (1 mL on each side) of Sunecos-200 solution (HA and AAs) were injected into the buccal mucosa four times at two-week intervals. The distance between the points of the injections was approximately 10 mm. The total number of injection points per side was 5. Cosmetic syringes (1 ml) and needles 30 G 4 mm were used for injection.
  Arms: Study group with intervention of Sunecos-200; injectable HA and AA solution

SUMMARY:
The goal of this clinical trial is to learn if drug containing non-crosslinked hyaluronic acid and amino acids solution (Sunecos-200) works to treat hyposalivation in adults. It will also learn about the safety of drug Sunecos-200. The main questions it aims to answer are:

* Does Sunecos-200 improve the saliva secretion and improve a life comfort?
* What medical problems do participants have when taking Sunecos-200? Researchers will compare drug containing non-crosslinked hyaluronic acid and amino acids solution (Sunecos-200) to a control group (without intervention) to see if drug Sunecos-200 works to treat hyposalivation.

Participants will:

* Take drug Sunecos-200 by into oral mucosa injection or nothing every two weeks for 4 times.
* Visit the clinic once every 2 weeks for checkups and tests
* Keep a diary of their symptoms after injection and fill out a primary and final questionary.

DETAILED DESCRIPTION:
Dry mouth is one of the most common complaints among patients, in both dental and general medicine practices, especially among the older population. Xerostomia (or dry mouth) is a medical term used to describe the subjective sensation of dry mouth that commonly occurs because of decreased salivary flow (hyposalivation). Although the two terms do not correspond to the same conditions and should not be used interchangeably, many physicians do so, since most patients with xerostomia also have hyposalivation.

Approximately 30% of the population complains on some degree of dry mouth. When it happens occasionally, during dehydration or stress, it is not a cause for concern. The situation is more serious if it happens more often, such as every day. It could also point to an underlying health condition. In untreated patients, hyposalivation increase their vulnerability to tooth decay, gingivitis and oral mucosa sensation. Dry mouth is related to pain, sometimes insomnia and psychological problems and results in deterioration of life well-being.

Saliva is produced by major salivary glands (MaSGs), the parotid, submandibular and sublingual glands and by circa 600 to 1,000 minor salivary glands (MiSGs) located in the submucosa layer in the oral cavity. MaSG contributed to 90% of total saliva secretions, whereas MiSG contributed to the remaining 10%. MiSGs are important for preventing the subjective sensation of dry mouth, since the saliva produced by these glands creates a lubricating micron-thick film that protects the oral mucosae. Furthermore, MiSGs play a key role in saliva production during sleep; therefore, reduced MiSG flow appears to be a cause of nocturnal dry mouth.

Saliva is a hypotonic solution composed of 98.5% water with 1% organic and 0.5% inorganic components. The organic and inorganic components of saliva are present in low concentrations, with some proteins synthetized in the gland (such as α-amylase) present in relatively high concentrations. Other organic components detected in saliva are vitamin C, maltase, urea, uric acid, lactase, hormones (testosterone, cortisol), albumin, creatinine, amino acids, mucin and immunoglobulins (IgA, IgG, IgM). Saliva α-amylase and lipase play a role in starch digestion and triglyceride decomposition. Salivary mucins lubricate intraoral structures and help to form a barrier against microbial invasion. Salivary immunoglobulins, especially secretory IgA (SIgA), play a key role in neutralizing toxins, agglutinating bacteria, and preventing their adhesion to mucosal surfaces.

By moistening the oral mucosa, saliva facilitates chewing, swallowing, and speech. Furthermore, a constant flow of saliva facilitates the mechanical removal of food debris and microorganisms and regulates the oral pH, protecting against acidic byproducts of bacterial metabolism. This buffering capacity is essential for maintaining a healthy oral microbiome and preventing demineralization of tooth enamel. Saliva also serves as a protective factor against infections because of its numerous organic components. People with dry mouth not only have trouble chewing and swallowing food but also have difficulty with tasting, speaking, and a reduced tolerance for dentures. Furthermore, xerostomia increases the risk of caries, periodontal disease, candidiasis, oral ulcers, and dysphagia, which can negatively impact nutritional status and quality of life.

There is wide variability in individual salivary flow rates. The average daily flow of whole saliva varies between 0.5 and 1.5 L. The accepted range for normal unstimulated salivary flow is above 0.1 ml/min. Any unstimulated flow rate below 0.1 ml/min is considered hypofunction. Stimulated saliva represents 80 to 90 % of daily salivary production, and the stimulated flow rate varies from 1 to 3 mL/minute.

Several studies have considered changes in saliva quantity and quality throughout the lifetime. No consensus has been reached on the decrease in the salivary flow rate with age. Despite this, recent research by Vandenberghe-Descamps et al revealed a 38.5% reduction in the resting salivary flow rate and 38.0% reduction of stimulated salivary flow rate in elderly subjects compared with young subjects. The cause of salivary flow decline has been connected to the loss of acinar cells; loss of secretory tissue and adiposity increase, as well as neurophysiological deterioration. Additionally, changes in saliva composition with age have been reported in some studies. Most notably, the mucin concentration decreases, which promotes the development of diseases of the oral mucosa and dry mouth.

Given the impact of reduced salivary flow on quality of life and oral health, assessing salivary function should be part of routine dental examinations, especially since saliva sampling is easy and noninvasive. The most advocated clinical method for diagnosing salivary gland dysfunction is to quantify unstimulated and stimulated whole saliva flow rates (sialometry). Recently, the Clinical Dry Mouth Score (CODS) was developed to objectively quantify clinical signs of decreased salivary flow. The CODS aims to provide a quick, easy, and objective method for assessing salivary gland function in a clinical setting. The CODS assesses dry mouth through clinical and visual examination of the oral cavity on the basis of several signs of dryness, such as frothy saliva, dry oral mucosa, and sticking of the mouth mirror to the tongue or cheek fold.

Despite the various etiological factors underlying xerostomia, the available treatment options do not differ on the basis of the cause and are predominantly symptomatic-except in cases of drug-induced xerostomia, where therapy involves discontinuation of the systemic medication.

Therapeutic strategies implemented to manage xerostomia, regardless of its etiology, have thus far failed to yield definitive or consistently effective outcomes.

ELIGIBILITY:
Inclusion Criteria:

* subjective feeling of dry mouth caused by a lack of saliva for at least 3 month,
* informed consent sing by patient,
* other complains including difficulty during eating, speaking or swallowing, taste disorders, trouble wearing dentures, the sensation that the tongue is stuck to the palate, bad breath and insomnia, feeling dry mouth at night, which made it difficult or impossible to sleep.

Exclusion Criteria:

* smoking,
* alkohol drinking,
* pregnancy,
* breast feeding,
* diabetes,
* immunosuppressive treatment,
* neoplastic diseases,
* Sjögren disease,
* active inflammation in the oral cavity,
* participation in other clinical trial in within the last 3 months,
* allergy or hipersensitivity to hyaluronic acid or amino acides,
* no planned hospital stay during the study

Ages: 38 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
Patient-reported pain connected with oral dryness using Visual Analog Scale (VAS) | Baseline
  The Visual Analogue Scale (VAS) assess the pain intensity on a scale from 0 to 10, where 0 indicates no pain; 1-3 - indicates mild pain; 4-6 - indicates moderate pain; 7-9 - indicates severe pain; and 10 - indicates unbearable pain.
Patient-reported pain connected with oral dryness using Visual Analog Scale (VAS) | 8 weeks following the baseline
  The Visual Analogue Scale (VAS) assess the pain intensity on a scale from 0 to 10, where 0 indicates no pain; 1-3 - indicates mild pain; 4-6 - indicates moderate pain; 7-9 - indicates severe pain; and 10 - indicates unbearable pain.
Improvement in patients-reported oral dryness score using an auctorial questioner | Baseline
  The auctorial questioner conteins 10 questions based on Xerostomia Inventory test. The 5 stages Likert scale is used for answer: 1-never, 2-rarely, 3-sometimes, 4-often, 5-always. The score 11-20 means mild dryness; 21-35 means moderate dryness; 36-50 severe dryness. The change of 5 points or more in the score is considered a clinically significant outcome, indicatig the success of treatment.
Improvement in patients-reported oral dryness score using an auctorial questioner | 8 weeks following the baseline.
  The auctorial questioner conteins 10 questions based on Xerostomia Inventory test. The 5 stages Likert scale is used for answer: 1-never, 2-rarely, 3-sometimes, 4-often, 5-always. The score 11-20 means mild dryness; 21-35 means moderate dryness; 36-50 severe dryness. The change of 5 points or more in the score is considered a clinically significant outcome, indicatig the success of treatment.

SECONDARY OUTCOMES:
Changes in unstimulated saliva before HA and AAs injections - mirror test | Baseline
  A "mirror test" evaluates unstimulated saliva flow. The examination checks the mobility of dental mirror on chick's mucous membrane. The results were described as movable or unmovable dental mirror.
Changes in unstimulated saliva after HA and AAs injections - mirror test. | 8 weeks following the baseline
  A "mirror test" evaluates unstimulated saliva flow. The examination checks the mobility of dental mirror on chick's mocus membrane. The results were described as movable or unmovable dental mirror.
Consistency changes in unstimulated saliva before HA and AAs injections. | Baseline
  To evaluate unstimulated saliva characteristic, a Saliva-Check Buffer GC test kit was used. The consistency of unstimulated saliva was assessed visually by the same dentist. The consistency was described as watery, sticky or frothy according to instruction of a Saliva-Check Buffer GC test kit.
Consistency changes in unstimulated saliva after HA and AAs injections. | 8 weeks following the baseline
  To evaluate unstimulated saliva characteristic, a Saliva-Check Buffer GC test kit was used. The consistency of unstimulated saliva was assessed visually by the same dentist. The consistency was described as watery, sticky or frothy according to instruction of a Saliva-Check Buffer GC test kit.
pH changes in unstimulated saliva before HA and AAs injections. | Baseline
  To evaluate unstimulated saliva characteristic, a Saliva-Check Buffer GC test kit was used.
  The pH measurement was performed by placing a pH test strip in a sample of unstimulated saliva for 10 s and comparing the results with the test chart included in the package. The samples were divided into strongly acidic (pH 5.0-5.8), moderately acidic (pH 6.0-6.6) and healthy saliva (pH 6.8-7.8) groups.
pH changes in unstimulated saliva after HA and AAs injections. | 8 weeks following the baseline
  To evaluate unstimulated saliva characteristic, a Saliva-Check Buffer GC test kit was used.
  The pH measurement was performed by placing a pH test strip in a sample of unstimulated saliva for 10 s and comparing the results with the test chart included in the package. The samples were divided into strongly acidic (pH 5.0-5.8), moderately acidic (pH 6.0-6.6) and healthy saliva (pH 6.8-7.8) groups.
Quantity of saliva changes in stimulated saliva before HA and AAs injections. | Baseline
  To evaluate stimulated saliva characteristic, a Saliva-Check Buffer GC test kit was used.
  The quantity test of stimulated saliva was performed. The patient was instructed to chew a piece of wax to stimulate saliva production. for 5 minutes. Saliva volume was measured by checking the ml markings on the container wall.
Quantity of saliva changes in stimulated saliva after HA and AAs injections. | 8 weeks following the baseline
  To evaluate stimulated saliva characteristic, a Saliva-Check Buffer GC test kit was used.
  The quantity test of stimulated saliva was performed. The patient was instructed to chew a piece of wax to stimulate saliva production. for 5 minutes. Saliva volume was measured by checking the ml markings on the container wall.
Buffering capacity changes in stimulated saliva before HA and AAs injections. | Baseline
  To evaluate stimulated saliva characteristic, a Saliva-Check Buffer GC test kit was used.
  The buffering capacity test of stimulated saliva was performed. The test strip included in the test kit was used to test buffering capacity. The result was calculated after 2 minutes according to the conversion table provided in the kit.
Buffering capacity changes in stimulated saliva after HA and AAs injections. | 8 weeks following the baseline
  To evaluate stimulated saliva characteristic, a Saliva-Check Buffer GC test kit was used.
  The buffering capacity test of stimulated saliva was performed. The test strip included in the test kit was used to test buffering capacity. The result was calculated after 2 minutes according to the conversion table provided in the kit.

CONTACTS AND LOCATIONS:
Overall Officials: Marzena Liliana Wyganowska, Professor, Study Director — Poznan University of Medical Sciences
Locations (1):
- Department of Periodontology and Oral Mucosa Diseases, Poznan University of Medical Sciences, Poznan, Greater Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underline the results reported in this clinical trial will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 month after publication of the main resultsand ending 5 years thereafter.
Access Criteria: Data will shared with researchers who provide a methodically sound proposal approved by the study sponsor. Request should be directed to wyganowska@ump.edu.pl or sklewinsteinbock@ump.edu.pl